CLINICAL TRIAL: NCT04201288
Title: Brief Acceptance-Based Retention Intervention for Newly Diagnosed HIV Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1908002504; R01MH119919 (NIH)
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: HIV/AIDS
Keywords: Medication adherence; Treatment adherence; HIV; Acceptance and Commitment Therapy; Retention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance-Based Behavior Therapy (ABBT) (Experimental): The 2-session ABBT will be delivered in person at session 1 and by telephone at session 2.
  Interventions: Behavioral: Acceptance-Based Behavior Therapy (ABBT)
- Enhanced-Treatment-as-Usual (ETAU) (Placebo Comparator): In addition to receiving treatment-as-usual at the clinic, ETAU participants will receive a 2-session program of HIV education.
  Interventions: Behavioral: Enhanced-Treatment-as-Usual (ETAU)

INTERVENTIONS:
Behavioral: Acceptance-Based Behavior Therapy (ABBT) — Acceptance-Based Behavior Therapy (ABBT) In the first session, the interventionist will introduce the concept of acceptance and its possible benefits in the context of life values and participant-identified barriers to retention in care. Interventionists will help participants identify potential challenges to acceptance, including disclosure concerns. At the second session, participants will practice acceptance-based coping skills and a behavioral plan will be developed to target barriers identified in the first session. These discussions will help the participant clarify how best to align their values with decisions on how to manage their HIV.
  Arms: Acceptance-Based Behavior Therapy (ABBT)
Behavioral: Enhanced-Treatment-as-Usual (ETAU) — ETAU will consist of two brief sessions lead by study interventionists, performed at the same times and by same methods as ABBT. Topics of education include safe sex practices, review of treatment options, and review of HIV-related indices of health.
  Arms: Enhanced-Treatment-as-Usual (ETAU)

SUMMARY:
The overall aim of this program of research is to test a newly developed intervention, Acceptance-Based Behavior Therapy (ABBT), to improve HIV patients' commitment to medical care.

The purpose of the proposed project is to establish the efficacy of ABBT and examine its mechanisms of action. To achieve the specific aims, the investigators will conduct a randomized clinical trial (n = 270), with two treatment arms: ABBT vs. an attention-matched HIV education control condition.

DETAILED DESCRIPTION:
Drop-out rates from medical clinics in the first months following linkage to HIV care are as high as 50%, with 31-46% of patients dropping out after the first visit. People Living with HIV (PLWH) who are not consistently retained in care are at risk for: delayed antiretroviral treatment (ART) initiation, reduced ART adherence, unsuppressed viremia, and mortality. Moreover, poor retention means effective ART cannot be leveraged to prevent further HIV transmission. The objective of this study is to conduct a fully powered, randomized controlled trial (RCT) to assess the efficacy of a brief, 2-session acceptance-based behavioral therapy (ABBT) intervention to enhance retention in HIV care.

The aims of this proposal are: (1) To test, in a 2-arm RCT, the efficacy of the ABBT intervention on retention in care and virologic suppression (primary outcomes); and, ART adherence, disclosure of HIV status, perceived social support, HIV stigmatization (secondary outcomes), relative to an Enhanced-Treatment-as-Usual condition; and, (2) To examine the degree to which retention in HIV care and virologic suppression are mediated by (a) increased HIV acceptance (and decreased HIV experiential avoidance) and (b) increased willingness to disclose HIV status. The sample will consist of 270 HIV patients who are new to care.

ELIGIBILITY:
Inclusion Criteria:

1. HIV+
2. ≥18 years old
3. Entering HIV medical care services for the first time (that is, not transferring HIV care from another location)
4. Able to speak and read English at the level to be able to complete the study procedures
5. Have telephone access.

Exclusion Criteria:

1. Cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Moitra, Ph.D., Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share data via the Research Data Center at the CDC's National Center for Health Statistics (NCHS).
Time Frame: Data will be shared upon the completion of the study and after summary data are published in a peer-reviewed journal. Consistent with NIMH guidelines, there will be no specific time limit regarding how long IPD are available.
Access Criteria: Request to access the data will be evaluated by the PI to ensure that they meet reasonable standards of scientific integrity.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred during routine intake at HIV clinics in Minneapolis, New Orleans, and Providence from December 2021 through March 2024.
Pre-assignment Details: Randomization was stratified by active substance use and depression severity.
Period: Overall Study
Arm/Group | Acceptance-Based Behavior Therapy (ABBT) | Enhanced-Treatment-as-Usual (ETAU)
Started | 20 | 16
Completed | 13 | 12
Not Completed | 7 | 4
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 5 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acceptance-Based Behavior Therapy (ABBT) | Enhanced-Treatment-as-Usual (ETAU) | Total
Number analyzed (Participants) | 20 | 16 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 16 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (8.4) | 32.8 (13.5) | 32.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 19 | 14 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 4 | 8
  White | 10 | 9 | 19
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 16 | 36
Addiction Severity Index [Count of Participants; unit: Participants] — Number of participants endorsing current (past month) non-prescribed substance use (opioids and/or stimulants).
  Participants | 4 | 2 | 6
AUDIT-C [Mean (Standard Deviation); unit: units on a scale] — Alcohol Use Disorders Identification Test - Concise (AUDIT-C) is a brief 3-item screener for hazardous alcohol use. A total score is calculated by summing the items, with a possible range of 0-12, with higher scores representing more hazardous alcohol use (worse outcome).
  units on a scale | 3.7 (2.6) | 3.8 (3.1) | 3.8 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Meeting Retention in HIV Medical Care Guidelines at 52 Weeks
Description: Objective data from participants' electronic health records will be obtained to examine how many medical appointments they attended in the past year at their HIV treatment clinic. Participants will be deemed as sufficiently retained if they attend at least 3 medical visits during this period.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Acceptance-Based Behavior Therapy (ABBT) | Enhanced-Treatment-as-Usual (ETAU)
Number analyzed (Participants) | 20 | 16
Participants | 20 | 16

2. Primary Outcome: Number of Participants Who Met HIV Virologic Suppression
Description: Objective data from participants' electronic health records will be obtained to examine their viral load, which is a blood-based measure of the amount of HIV viruses in the person's body. If participants are not currently retained in medical care and blood sample results are not available in their electronic health record, they will submit 1-3ml of blood at each assessment through the study's research phlebotomist. A viral load that measures as "undetectable" (i.e., fewer than 200 copies of HIV per millilitre of blood) will represent virologic suppression, which is a positive indication of HIV health.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Acceptance-Based Behavior Therapy (ABBT) | Enhanced-Treatment-as-Usual (ETAU)
Number analyzed (Participants) | 20 | 16
Participants | 20 | 14

3. Secondary Outcome: Self-Rating Scale Item (SRSI) - Antiretroviral Treatment Adherence
Description: Self-report data of participants' HIV antiretroviral treatment adherence will be obtained with the SRSI. Scores range from 0 to 5, which correspond to "very poor" to "excellent" medication adherence.
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acceptance-Based Behavior Therapy (ABBT) | Enhanced-Treatment-as-Usual (ETAU)
Number analyzed (Participants) | 13 | 12
score on a scale | 4.5 (0.7) | 4.6 (0.7)

4. Secondary Outcome: Brief HIV Disclosure Scale (BHD)
Description: The BHD HIV disclosure scale will be used to assess for willingness to make informed disclosure and for actual disclosure of HIV status. Scores range from 8-32, with higher scores indicating increased willingness to disclose.
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance-Based Behavior Therapy (ABBT) | Enhanced-Treatment-as-Usual (ETAU)
Number analyzed (Participants) | 13 | 12
units on a scale | 21.3 (3.2) | 22.1 (4.2)

5. Secondary Outcome: The Multidimensional Scale of Perceived Social Support (MSPSS)
Description: The MSPSS will be used to measure perceived social support. Scores range from 1-84, with higher scores indicating greater perceived social support.
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance-Based Behavior Therapy (ABBT) | Enhanced-Treatment-as-Usual (ETAU)
Number analyzed (Participants) | 13 | 12
units on a scale | 5.8 (0.7) | 5.3 (0.9)

6. Secondary Outcome: HIV Stigma Scale (HSS)
Description: The HSS will be used to measure self-reported experiences, fear, and perception of stigmatization due to being HIV+. Scores range from 6-24, with lower scores indicating less fear or concern about stigmatization.
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance-Based Behavior Therapy (ABBT) | Enhanced-Treatment-as-Usual (ETAU)
Number analyzed (Participants) | 13 | 12
units on a scale | 19.5 (4.5) | 21.1 (5.0)

ADVERSE EVENTS:
Time Frame: Duration of the study, which was 4 years.
Arm/Group | Acceptance-Based Behavior Therapy (ABBT) | Enhanced-Treatment-as-Usual (ETAU)
All-Cause Mortality (participants affected / at risk) | 1/20 | 1/16
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/16
Other Adverse Events (participants affected / at risk) | 0/20 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT04201288/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT04201288/SAP_001.pdf
  • Informed Consent Form (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT04201288/ICF_002.pdf